CLINICAL TRIAL: NCT03977012
Title: Neuroimaging Study on the Effect of Transdermal Buprenorphine in Complex Regional Pain Syndrome(CRPS) Patients With Chronic Lower Back Pain: A Pilot Study
Brief Title: Neuroimaging Study on the Effect of Transdermal Buprenorphine in Complex Regional Pain Syndrome Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Hee Choi, Associate Professor, Seoul National University Hospital
Other Study IDs: NOR17-KR-IIT
Record Dates: First submitted 2019-05-23; First posted 2019-06-06 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Complex Regional Pain Syndromes
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Buprenorphine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with CRPS Type I: Patients diagnosed with Complex Regional Pain Syndrome Type I who are anticipated to recieve a 8 weeks regime of buprenorphine as a part of routine medical care.
  -drug name: norspan patch 5~20 mcg dosage form: patch frequency: every weeks duration: 8 weeks
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — 5~20 mcg
  Other Names: norspan patch

SUMMARY:
In the present study, we aim to investigate the effect of buprenorphine on neuroinflammation in patients with complex regional pain syndrome, using [11C]-(R)-PK11195 PET.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with complex regional pain syndrome Type I (Budapest Criteria) and persistent back pain (VAS ≥ 4).
2. Patients who can stop benzodiazepine treatment 2 weeks before study
3. Patients who initially decided to use buprenorphine according to clinical judgment
4. Patients who are able to understand the purpose and procedure of the study

Exclusion Criteria:

1. Patients with an impaired cognitive function such as psychosis, dementia, or mental retardation
2. Patients with neurologic disease, cerebrovascular disease, history of brain tumor, history of severe head trauma, history of convulsive disease
3. Patients with cardiovascular disease, liver, respiratory or renal dysfunction
4. Patients with biliary disease
5. Patients who could not undergo the PET/magnetic resonance imaging (MRI) process.
6. Patients who have a risk of suicide or show aggressive behavior
7. Patients who have drug dependence (DSM-IV criteria) or history (past 6 months or older)
8. Employees of researchers or clinical research institutes
9. Patients with hypersensitivity or contraindication to buprenorphine

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients diagnosed with complex regional pain syndrome Type I (Budapest Criteria)
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-06-11 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Changes in neuroinflammation | baseline, 8 weeks
  [11C]-(R)-PK11195 PET distribution volume ratio (DVR)

SECONDARY OUTCOMES:
Morphine equivalent | baseline, 8 weeks
  narcotic analgesic dosage
Physical test(1) | baseline, 8 weeks
  blood test
Physical test(2) | baseline, 8 weeks
  urine test
Physical test(3) | baseline, 8 weeks
  Electrocardiogram(ECG) test (pulse rate)
Physical test(4) | baseline, 8 weeks
  pulse measurement
Physical test(5) | baseline, 8 weeks
  blood pressure measurement
Self-reported questionnaire(1) | baseline, 8 weeks
  Beck Depression Index(BDI)/ total score: 0~63, The higher the score, the more depressed
Self-reported questionnaire(2) | baseline, 8 weeks
  Beck Anxiety Index(BAI)/ total score: 0~63, The higher the score, the more anxiety
Self-reported questionnaire(3) | baseline, 8 weeks
  Short Form McGill Pain Questionnaire(SF-MPQ)/ 'a' subscale score: 0~45, The higher the score, the more painful/ 'b' subscale score, 0~10, The higher the score, the more painful/ 'c' subscale score, 0~5, The higher the score, the more painful
Self-reported questionnaire(4) | baseline, 8 weeks
  Pain Catastrophizing Scale/ total score: 0~52, The higher the score, the more pain Catastrophizing

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No